CLINICAL TRIAL: NCT06871436
Title: Telerehabilitation as a Follow-up Modality for Obese People After Returning Home Following Hospitalization
Brief Title: Telerehabilitation as Follow-up for Obesity
Acronym: OPaCTe
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de l'Obesite Bernard Descottes (Other)
Collaborators: Limoges University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N° 2024-A02428-39
Record Dates: First submitted 2025-02-10; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Obese Patients
Keywords: Telerehabilitation; Obesity; Adults; Physical Exercise; Mindsets
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Supervised Telerehabilitation (Experimental): Participants will have access to the Follow SURG application to monitor their health at home. In addition, participants will be asked to wear the activity wristband daily (except when sleeping) and to download the GARMIN Connect app on their smartphone to update their physical activity data. They will participate in telerehabilitation sessions with a professional via videoconference using the AXOMOVE telehealth application.
  These sessions will take place three times a week, for 60 minutes, from 12pm to 13pm and 5pm to 6pm on Mondays, Wednesdays and Fridays. Each telerehabilitation group will follow these sessions live. Telerehabilitation sessions include a 10-minute warm-up, 40 minutes of circuit training, 5 minutes of stretching and 5 minutes of discussion with the professional.
  Interventions: Other: Aerobic Exercice and muscular reinforcement
- Unsupervised Physical Activity Videos (Experimental): Participants will be able to use the Follow SURG application to monitor their health at home. In terms of accessibility, this will be comprehensive, with access to informative content proposed by paramedical professionals such as psychomotricians, dieticians and psychologists, as well as content made available in the current COBD follow-up. In addition, participants will be asked to wear the activity wristband on a daily basis (except when sleeping) and to download the GARMIN Connect application onto their smartphone in order to update their PA data. Participants will be asked to carry out APA sessions 3 times a week, using videos produced in advance by a professional. Videos will include 10 min of warm-up, 40 min of circuit training (following the same modalities as those defined in the "Telerehabilitation" section) and 10 min of stretching.
  Interventions: Other: Aerobic Exercice and muscular reinforcement
- Contrôle Group (No Intervention): Participants will be able to use the Follow SURG application to monitor their health at home. Access to the Follow SURG application will be restricted to informative content provided by paramedical professionals such as psychomotricians, dieticians and psychologists. In addition, participants will be asked to wear the activity wristband on a daily basis (except when sleeping) and to download the GARMIN Connect app on their smartphone in order to update their physical activity data. In addition, reminders to practice physical activity will be provided on the Follow SURG app 3 times a week.

INTERVENTIONS:
Other: Aerobic Exercice and muscular reinforcement — Aerobic exercise and muscle strengthening to increase weekly physical activity at moderate and vigorous intensities
  Other Names: Physical activity; Exercise; muscular reinforcement
  Arms: Supervised Telerehabilitation; Unsupervised Physical Activity Videos

SUMMARY:
The goal of this experimental study is to observed the impact of telerehabilitation modalities in obese patient after a hospitalization on physical intensity at home (MVPA). The secondary aim is to observe the evolution of clinical parameters such as anthropometric data, adherence and psychological state.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 years old)
* BMI > 35 or 30 Kg/m2 in case of concomitant comorbidity
* Authorization to practice physical activity for participants over 30 years old by means of a cardiac assessment and an ECG less than 6 months old carried out by a cardiologist. As part of the COBD treatment, the ECG is either: integrated into the patient file before hospitalization if the patient has seen his cardiologist staff. Either the ECG is provided in the file or carried out and analyzed by the center's cardiologist (Dr Rouffaud). The latter then authorizes or not the practice of PA.
* Complete 3-week stay in an obesity center
* Availability of equipment suitable for telerehabilitation at home
* Having given informed consent for participation in the study

Exclusion Criteria:

* Medical contraindication to PA practice defined by a doctor
* Participation in a concomitant research protocol
* For women of childbearing age, they will be informed that in the event of pregnancy occurring during participation in the research, they will not be able to continue the protocol and will withdraw from the research
* Refusal to participate in the research protocol
* Patient on weekday stay (< 3 weeks)
* Psychiatric/psychological disorder limiting the expression of consent
* Persons under legal protection or unable to express their consent
* Inability to participate in any of the 18 Telerehabilitation sessions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-04-07 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-08-07 (Estimated)

PRIMARY OUTCOMES:
MVPA | Up to 8 months
  Time (min/s) of physical activity at moderate and/or vigorous intensity. This is done with a trivial accelerometer and measures with an equation (Garmin) the MVPA practice time over a week and gives a value in minutes per week. It enables us to understand whether or not a participant is achieving the recommended level of physical activity (150 min/week at moderate or vigorous intensity).
MVPA | Up to 8 months
  This questionnaire by Craig et al (2003) consists of 27 questions divided into 5 parts. In each part, the participant is asked to quantify the amount of time in minutes/hours/days spent in PA. The first part comprises questions 1 to 7 and covers all physical activity practised in a professional context. The second part, questions 8 to 13, covers physical activity related to daily commuting (walking, cycling, driving, etc.) (to work, to the stores, etc.). The third part comprises questions 14 to 19 and covers activities related to housework, home maintenance, time spent with family, etc. The fourth part, questions 20 to 25, deals with physical activity related to leisure, sport and free time. Finally, the fifth section includes questions 26 to 27 and covers time spent sitting or lying down during the day.

SECONDARY OUTCOMES:
Weight | Up to 8 months
  weight of participants in kilograms
Walking Distance | Up to 8 months
  The walking test will be performed in a corridor delimited by two markers spaced 30 meters apart, following international recommendations (Baillot, Baillargeon, Brown & Langlois, 2015). The distance is calculated using markers placed on the ground at the end of the test. In addition, dyspnea and perception of effort were measured at the end of the test using the modified BORG scale (0 representing a dyspneic state or non-existent difficulty in exertion and 10 a dyspneic state or perception of maximum effort).
Effort perception and dyspnea | Up to 8 months
  Assessment of perceived exertion and dyspnoea after exercise using the modified Borg scale. This scale ranges from 1 to 10. A score close to 1 shows a perception of effort and a feeling of weak dyspnea. Conversely, the higher the score, the more difficult the effort is perceived.
Lower limb strength | Up to 8 months
  The chair stand-up test will be implemented with a chair placed against a wall. The subject must stand up and sit down as many times as possible from their chair in 30 seconds, without leaning against the backrest and using their hands. This version will be applied since its reliability and reproducibility is greater in subjects whose average age is less than 65 years (Orange et al., 2018).
Adhesion to telerehabilitation | Up to 6 weeks
  There will be 18 sessions to do in total and the percentage of participation will be estimated from this number of sessions.
Intensity of sessions | Up to 6 weeks
  Intensity of sessions measured with Garmin wristband to obtain reserve heart rate during sessions. Reserve heart rate will be measured with the formula : Max Heart Rate - Rest Heat Rate. Participants need to train at 60% of RHR.
Digital tool acceptance | up to 6 weeks
  The Technology Acceptance Model (TAM) questionnaire was developed in its first version by Davis (1989). The version used is a French translation by Hayotte et al., (2020). It consists of 16 items and follows a Likert scale ranging from 1 to 7 (respectively from "strongly disagree" to "strongly agree"). It measures the perception of a digital tool by subjects. This questionnaire will be used twice, first to measure the acceptability of the digital tool used during the first meeting with patients, then secondly for the acceptance of the digital tool at the end of the various remote sessions.
sedentary lifestyle | Up to 8 months
  measured with the IPAQ questionnaire. This questionnaire by Craig et al (2003) consists of 27 questions divided into 5 parts. In each part, the participant is asked to quantify the amount of time in minutes/hours/days spent in PA. The first part comprises questions 1 to 7 and covers all physical activity practised in a professional context. The second part, questions 8 to 13, covers physical activity related to daily commuting (walking, cycling, driving, etc.) (to work, to the stores, etc.). The third part comprises questions 14 to 19 and covers activities related to housework, home maintenance, time spent with family, etc. The fourth part, questions 20 to 25, deals with physical activity related to leisure, sport and free time. Finally, the fifth section includes questions 26 to 27 and covers time spent sitting or lying down during the day.
Self Esteem | Up to 8 months
  The "self-esteem" test is a self-questionnaire created by Rosenberg (1968) whose French version is that of Vallières and Vallerand (1990). The test consists of 10 "Likert" type items with reverse item coding. This scale is based on 4 choices organized from 1 to 4 ranging respectively from "completely disagree" to "completely agree".
Body perception | Up to 8 months
  Body perception questionnaire with figure rating scale. The "Figure Rating Scale" test was developed by Stukard et al. (1983). This test measures the difference between the perceived and ideal body shape of obese people. This test consists of 9 figures numbered from 1 to 9. First, the participant must circle the figure representing the "perceived" physique (their situation at a given time) and then circle the figure representing the "ideal" physique to be achieved. An indicator is then calculated by taking the difference between the ideal score and the perceived score.
Quality of living | up to 8 months
  Measuring quality of life with the SF-36 questionnaire. The SF-36 is a quality of life questionnaire validated in France by Leplege et al. (1998). This test consists of 36 questions and is based on two dimensions of quality of life: physical and mental health. The questions cover physical mobility, limitations in the practice of daily activities, bodily pain, general health, vitality, bio-psycho-social approach and mental health. Standardized scores range from 0 (poor health) to 100 (good health).
implicit beliefs about weight loss | Up to 8 months
  Questionnaire to measure implicit beliefs related to the ability to regulate one's weight. This scale, proposed by Brunette (2010) is an adaptation of an instrument initially created by Dweck & Leggett (1998). Since no version translated into French existed in the literature, we will instead carry out a double translation of the original instrument using two bilingual people. Three researchers who had previously worked in the field of obesity agreed on the final version in French. This questionnaire consists of 6 items following a Likert scale ranging from 1 "Always" to 6 "Never" and measuring the subjects' relative beliefs regarding their ability to regulate their body mass.
Self-efficacy linked to physical activity | Up to 8 months
  Sense of self-efficacy related to physical activity measured by a 2-subscale questionnaire. This questionnaire is the French version of the "Exercice Confidence Survey" (Sallis, 1996) validated by Eeckhout et al. (2012). It consists of 12 items following a Likert scale ranging from 1 "I know I can't" to 5 "I know I can". It is divided into two sub-dimensions, namely: measurement of adherence to PA comprising 8 items (1, 2, 3, 4, 5, 6, 7, 8) and measurement of constraints to PA practice with 4 items (9, 10, 11, 12).
Motivation to physical activity | Up to 8 months
  Measuring the nature of motivation for physical activity with the EMAPS questionnaire. This French questionnaire consists of 18 items on a Likert scale ranging from 1 "Does not correspond at all" to 7 "Corresponds very strongly". It aims to measure the different types of motivation for PA in subjects suffering from chronic pathologies according to the continuum proposed by Deci and Ryan (2002). This scale is divided into 6 sub-dimensions, each measuring a specific component of motivation, each comprising 3 items: intrinsic (1, 6, 11), integrated extrinsic (7, 10, 13), identified extrinsic (4, 12, 16), introjected extrinsic (3, 14, 18), external regulation extrinsic (9, 15, 17) and amotivation (2, 5, 8).
Size | Up to 8 months
  Size measured in Centimeters
Fat Mass | Up to 8 months
  fat mass (%) measured in the morning on an empty stomach (whenever possible) using a Tanita impedance meter (MC-780MA P, Tanita Europe B.V., Amsterdam, The Netherlands).
Fat Free Mass | Up to 8 months
  fat free mass (Kg) measured in the morning on an empty stomach (whenever possible) using a Tanita impedance meter (MC-780MA P, Tanita Europe B.V., Amsterdam, The Netherlands).
Waist circumference | Up to 8 months
  waist circumference (cm) measured by a Doctor according to a standardized protocol.
Intensity of sessions | Up to 6 weeks
  Participants will be asked to report their feelings of exertion and sensation of dyspnea during the sessions. Assessment of perceived exertion and dyspnoea after exercise using the modified Borg scale. This scale ranges from 1 to 10. A score close to 1 shows a perception of effort and a feeling of weak dyspnea. Conversely, the higher the score, the more difficult the effort is perceived.
Body dissatisfaction | Up to 8 months
  The body dissatisfaction test comes from the Eating Disorders Inventory-II developed by Garner et al. (1983), the French version of which is the work of Criquillon-doublet et al. (1995). This test measures personal dissatisfaction with the subjects' body segments or parts. This test consists of 9 items on a 6-level Likert scale ranging from: 1 "never" to 6 "always".

CONTACTS AND LOCATIONS:
Overall Officials: Claudine VASSEUR, Coordinating doctor, Principal Investigator — Centre de l'Obesite Bernard Descottes
Locations (1):
- Bernard Descottes Obesity Center, Saint-Yrieix-la-Perche, France

IPD SHARING:
Plan to Share IPD: Undecided